CLINICAL TRIAL: NCT03720938
Title: A Digital Movement in the World of Inactive Children: Outcomes of Playing Active Video Games in a Pilot Randomized Trial
Brief Title: Effects of Active Video Games in Physically Inactive Children
Acronym: AVGAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Dilsad Coknaz, Associate Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012.16.02.545
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Self-Perception; Body Weight
Keywords: inactive children; active video games; physical fitness; self-perception; enjoyment; obesity
MeSH Terms: conditions — Body Weight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Physically inactive children who did not play AVGs.
- Intervention Group (Experimental): Physically inactive children who played alternately Nintendo Wii® active video games for 50-60 min, 3 days a week, 12 weeks, in laboratory environment.
  Interventions: Other: Active Video Games

INTERVENTIONS:
Other: Active Video Games — Nintendo Wii® AVGs from sports, balance, aerobics, resort and training categories.
  Arms: Intervention Group

SUMMARY:
Inactivity was reported to be high in children and considered to be the fourth common cause of death in all ages. The reason for children is usually the increasing indoor use of sedentary screen time. Active Video Games (AVG) have recently been introduced for decreasing the sedentary time for children and directing them to physical activity (PA) at home.The aim of this study is to show the quantitative effect of games on physical fitness parameters like weight, body mass index (BMI) and fat ratio (FR). The study also aims at the factors for motivation or continuance of the games as self-perception and enjoyment levels together with qualitative effects of games on satisfaction and attitude changes in inactive children.

DETAILED DESCRIPTION:
Research related a causal association between inactivity, low esteem, and excess weight for children. For this reason, academic performance decreases and obesity associated diseases such as hypertension, diabetes, coronary heart diseases, depression, and cancer might ensue. Children usually do not prefer to perform outdoor PA due to several causes including low sense of self perception.

So far studies have shown an almost equivalent energy spent through AVGs to the physical activity of moderate intensity. Games have been previously demonstrated to prevent excess weight. There were no studies of AVG in children with varying weights, inactivity and technology preoccupation. Similarly, no qualitative research of AVG in children exploring enjoyment levels and attitude changes were encountered.

Thus, the investigators aim to find the quantitative effect of AVG on physical fitness parameters like weight, BMI and FR. Other aims are studying factors for motivation or continuance of the games as well as the feelings and perspectives of the participant children's parents for the games.

ELIGIBILITY:
Inclusion Criteria:

1. Being 8-13 years old
2. Being preoccupied with technology
3. Being physically inactive

Exclusion Criteria:

1. Having circulatory, respiratory and musculoskeletal disease
2. Having neuropsychiatric diseases
3. History of syncope or seizures
4. History of exercise induced anaphylaxis
5. Morbid obesity
6. Short stature

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dilsad Coknaz, Principal Investigator — Abant Izzet Baysal University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohl HW 3rd, Craig CL, Lambert EV, Inoue S, Alkandari JR, Leetongin G, Kahlmeier S; Lancet Physical Activity Series Working Group. The pandemic of physical inactivity: global action for public health. Lancet. 2012 Jul 21;380(9838):294-305. doi: 10.1016/S0140-6736(12)60898-8. PMID 22818941
- [Background] Booth FW, Roberts CK, Laye MJ. Lack of exercise is a major cause of chronic diseases. Compr Physiol. 2012 Apr;2(2):1143-211. doi: 10.1002/cphy.c110025. PMID 23798298
- [Background] Maddison R, Foley L, Mhurchu CN, Jull A, Jiang Y, Prapavessis H, Rodgers A, Vander Hoorn S, Hohepa M, Schaaf D. Feasibility, design and conduct of a pragmatic randomized controlled trial to reduce overweight and obesity in children: The electronic games to aid motivation to exercise (eGAME) study. BMC Public Health. 2009 May 19;9:146. doi: 10.1186/1471-2458-9-146. PMID 19450288
- [Background] Martins C, Morgan L, Truby H. A review of the effects of exercise on appetite regulation: an obesity perspective. Int J Obes (Lond). 2008 Sep;32(9):1337-47. doi: 10.1038/ijo.2008.98. Epub 2008 Jul 8. PMID 18607378
- [Derived] Coknaz D, Mirzeoglu AD, Atasoy HI, Alkoy S, Coknaz H, Goral K. A digital movement in the world of inactive children: favourable outcomes of playing active video games in a pilot randomized trial. Eur J Pediatr. 2019 Oct;178(10):1567-1576. doi: 10.1007/s00431-019-03457-x. Epub 2019 Aug 30. PMID 31471690
- See also: Global Strategy on Diet, Physical Activity and Health — http://www.who.int/dietphysicalactivity/physical_activity_intensity/en/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four primary public schools among 14 in the central schools of Bolu region were randomly selected. In January to February of year 2013, all children (n=1300) from grades III,IV,V and VI were given froms for participation.Children positively responded to informed consent forms (n=918) were accepted as eligible for the study.
Pre-assignment Details: The discrepancy between the enrolled (918) and assigned (n=106) numbers of children could be attributed to strict "inclusion" and "exclusion" criteria, and particularly to dropped out children due to technological preoocupation and physical inactivity as well as problems interfering physical activity and self-perception.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 242 | 676
Completed | 53 | 53
Not Completed | 189 | 623

BASELINE CHARACTERISTICS:
Population: Techologically preoccupation and low physical activity
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.31 (1.15) | 9.62 (1.02) | 9.96 (1.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
  Male | 22 | 24 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 53 | 53 | 106
Techonology pre-occupation and physical inactivity [Number; unit: participants] — "Technology preoccupied" children were determined if children were using the computer for activities other than homework, for at least 7 h or more in a week, watching television for 3 h or more in a day, playing video games for 5 h or more in a week in addition to the parental definition of the children as preoccupied with technology.
  Similarly, "physically inactive" children were defined as having activity scores less than 1.56 by Ekelund Criteria. Activity scores were calculated by dividing daily energy consumptions by basal metabolic rates described previously methods.
  participants | 53 | 53 | 106

OUTCOME MEASURES:

1. Primary Outcome: Weight in Kilograms
Description: Weight measured to the nearest 0.01 kg by Seca 767 scale. The first before the games, the second after the games.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Control Group: Physically inactive children who did not play AVGs.
  Active Video Games: Nintendo Wii® AVGs from sports, balance, aerobics, resort and training categories.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
kg
  At the beginning of games | 34.29 (8.46) | 33.65 (9.39)
  At the end of the games | 36.19 (9.04) | 34.18 (9.58)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable weight; Test type: Superiority — A sample size of 26 children per group was needed with the assumption of Cohen's d = 0.8, the alpha error of 0.05 and a power of 80%; p = 0.001, ANCOVA — The outcomes of weight was tested for any difference between groups by covariate analysis (ANCOVA) adjusted for the weight at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable weight; Test type: Other; p = 0.0002535, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted for cluster effect, and small sample sizes in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable weight; Test type: Superiority; p = 0.000397, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted by Satterthwaite's degrees of freedom method for cluster effect, and small sample sizes in addition to baseline value and age

2. Primary Outcome: Weight z Score
Description: Weight measured to the nearest 0.01 kg by Seca 767 scale. Z scores were calculated using national data for Turkish children. The first before the games, the second after the games. Positive z-scores indicates the number of standard deviations of the child above the mean of the population of the same age, whereas negative z-scores indicates the number of standard deviations of the child below the mean of the population of the same age.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
units on a scale
  At the beginning of games | -0.22 (1.05) | 0.13 (1.23)
  At the end of the games | 0.06 (1.02) | 0.23 (1.23)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable weight z scores; Test type: Superiority; p = 0.005, ANCOVA — The outcome of weight z score was tested for any difference between groups by covariate analysis (ANCOVA) adjusted for the weight at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable weight z score; Test type: Superiority; p = 0.002, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality. Adjusted by Satterthwaite's degrees of freedom correction method for cluster effect, and small sample sizes in addition to baseline value and age; Test type: Superiority; p = 0.00386, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

3. Primary Outcome: BMI Calculated as "Weight (kg) / Height (m^2)"
Description: Body Mass Index calculation of both groups before the games and after the games.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: kg/ m^2
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
kg/ m^2
  At the beginning of games | 18.20 (3.29) | 17.97 (3.34)
  At the end of the games | 18.86 (3.57) | 17.64 (3.36)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable body mass index; Test type: Superiority; p = 0.000, ANCOVA — The outcomes of weight was tested for any difference between groups by covariate analysis (ANCOVA) adjusted for the body mass index at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable body mass index; Test type: Superiority; p = 0.00000306, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality. Adjusted for cluster effect, and small sample sizes, baseline value and age; Satterthwaite's correction method for denominator degrees of freedom
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable body mass index; Test type: Superiority; p = 0.00000367, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

4. Primary Outcome: BMI z Score
Description: Weight and height were measured to the nearest 0.01 kg (Seca 767) and 0.1 cm (Seca 220). BMI Z-scores were calculated using national data for Turkish children derived from values obtained from calculations with Quetelet index. The first before the games, the second after the games. Positive BMI z-scores indicates the number of standard deviations of the child above the mean of the population of the same age, whereas negative z-scores indicates the number of standard deviations of the child below the mean of the population of the same age.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
units on a scale
  At the beginning of games | 0.06 (1.15) | 0.13 (1.30)
  At the end of the games | 0.27 (1.17) | 0.00 (1.31)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable body mass index z score; Test type: Superiority; p = 0.000, ANCOVA — The outcome of body mass index z score was tested for any difference between groups by covariate analysis (ANCOVA) adjusted for the body mass index z score at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable body mass index z score; Test type: Superiority; p = 0.0001402, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable body index z score; Test type: Superiority; p = 0.000235, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

5. Primary Outcome: Body Fat Percentage as Determined by Siri Formula From Skinfold Thicknesses
Description: The biceps, triceps, suprailiac and subscapular regions skinfold thicknesses were measured by Holtain caliper at the beginning of and after the games. Durnin-Womersley formula was used to calculate body densities. Then fat ratio of whole body was derived from the Siri equation by integrating body densities obtained by Durnin-Womersley formula.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
percentage of fat
  At the beginning of games | 25.43 (6.78) | 24.54 (7.14)
  At the end of the games | 24.62 (7.83) | 22.37 (6.68)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable fat ratio; Test type: Superiority; p = 0.259, ANCOVA — The outcomes of fat ratio was tested for any difference between groups by covariate analysis (ANCOVA) adjusted for the fat ratio at baseline and confounding variable age; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable fat ratio; Test type: Superiority; p = 0.220, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable fat ratio; Test type: Superiority; p = 0.250006, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

6. Secondary Outcome: Visual Reaction Times of Dominant Hand by Newtest 1000 Timer
Description: Determination of visual reaction times after games in intervention groups, and control groups. First before the games, second after the games.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
seconds
  At the beginning of games | 0.269 (0.055) | 0.263 (0.067)
  At the end of the games | 0.269 (0.075) | 0.233 (0.040)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable visual reaction time; Test type: Superiority; p = 0.000, ANCOVA — The outcome of visual reaction time was tested for any difference between groups by covariate analysis; Adjusted for the weight at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; The outcome of visual reaction time was tested for any difference between groups by linear mixed-effects model analysis; Test type: Superiority — Adjusted for the weight at baseline and confounding variable age; p = 0.00001196, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable visual reaction time; Test type: Superiority; p = 0.0000282‬, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

7. Secondary Outcome: Visual Reaction Times of Non-dominant Hand by Newtest 1000 Timer
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
seconds
  At the beginning of games | 0.284 (0.058) | 0.282 (0.083)
  At the end of the games | 0.282 (0.076) | 0.240 (0.045)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable visual reaction time of non-dominant hand; Test type: Superiority; p = 0.000, ANCOVA — The outcome of visual reaction time of non-dominant hand was tested for any difference between groups; Adjusted for the visual reaction time of non-dominant hand at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.00000009, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 000000055, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

8. Secondary Outcome: Auditory Reaction Time of Dominant Hand by Newtest 1000 Timer
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
seconds
  At the beginning of games | 0.314 (0.071) | 0.285 (0.079)
  At the end of the games | 0.289 (0.079) | 0.243 (0.053)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable auditory reaction time of dominant hand; Test type: Superiority; p = 0.000, ANCOVA — The outcomes of auditory reaction time of dominant hand was tested for any difference between groups by covariate analysis; Adjusted for the auditory reaction time of dominant hand at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.00001633, Linear mixed-effects model — The outcomes of auditory reaction time of dominant hand was tested for any difference between groups by linear mixed-effects analysis; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0000367, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

9. Secondary Outcome: Auditory Reaction Time of Non-dominant Hand by Newtest 1000 Timer
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
seconds
  At the beginning of games | 0.321 (0.074) | 0.294 (0.086)
  At the end of the games | 0.293 (0.080) | 0.264 (0.049)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable auditory reaction time of non-dominant hand; Test type: Superiority; p = 0.008, ANCOVA — The outcomes of auditory reaction time of non-dominant hand was tested for any difference between groups by covariate analysis; Adjusted for the auditory reaction time of non-dominant hand at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.006, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.006602, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

10. Secondary Outcome: Self-Perception of Sports Competence Assessed by Children and Youth Physical Self-perception Profile (CY-PSPP)
Description: The scale "Children and Youth Physical Self Perception Profile (CY-PSPP)" assessed the children's self-percetion about sports competence subscale in both groups at the beginning and at the end of protocol. The subscale was assessed by 6 questions with four ordinal levels (1-4) of response. Minimum and maximum total scores change between 6 to 24 for the subscale. Higher scores mean a better score.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
score on a scale
  At the beginning of games | 17.11 (2.59) | 16.11 (2.35)
  At the end of the games | 18.79 (2.95) | 17.73 (3.63)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable self-perception of sports competence; Test type: Superiority; p = 0.615648, ANCOVA — The outcome of self-perception for sports competence was tested for any difference between groups by covariate analysis; Adjusted for self-perception for sports competence at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; The outcome of self-perception for sports competence was tested for any difference between groups by linear mixed-effects model analysis; Test type: Superiority; p = 0.608, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.60938, Linear mixed-effects model — The outcome of self-perception for sports competence was tested for any difference between groups by linear mixed-effects model analysis; [statistical method as in outcome 1, analysis 3]

11. Secondary Outcome: Self-perception of Physical Condition Competence Assessed by Children and Youth Physical Self-perception Profile (CY-PSPP)
Description: The scale "Children and Youth Physical Self Perception Profile (CY-PSPP)" assessed the children's self-percetion about physical condition competence subscale in both groups at the beginning and at the end of protocol. The subscale was assessed by 6 questions with four ordinal levels (1-4) of response. Minimum and maximum total scores change between 6 to 24 for the subscale. Higher scores mean a better score.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
score on a scale | 18.15 (3.08) | 17.52 (2.78)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable self-perception of physical condition competence; Test type: Superiority; p = 0.094, ANCOVA — The outcome of self-perception for physical condition competence was tested for any difference between groups by covariate analysis; Adjusted for self-perception for physical condition competence at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.085, Linear mixed effects model — The outcome of self-perception for physical condition competence was tested for any difference between groups by linear mixed-effects model analysis; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.08818, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

12. Secondary Outcome: Self-perception of Strength Competence Assessed by Children and Youth Physical Self-perception Profile (CY-PSPP)
Description: The scale "Children and Youth Physical Self Perception Profile (CY-PSPP)" assessed the children's self-percetion about strength competence subscale in both groups at the beginning and at the end of protocol. The subscale was assessed by 6 questions with four ordinal levels (1-4) of response. Minimum and maximum total scores change between 6 to 24 for the subscale. Higher scores mean a better score.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
score on a scale
  At the beginning of games | 17.03 (3.05) | 16.35 (3.24)
  At the end of the games | 19.24 (3.27) | 17.49 (3.66)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable self-perception of strength competence; Test type: Superiority; p = 0.058102, ANCOVA — The outcome of self-perception for strength competence was tested for any difference between groups by covariate analysis; Adjusted for self-perception for strength competence at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.051, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0534, Linear mixed-effects model — The outcome of self-perception for strength competence was tested for any difference between groups by linear mixed-effects model analysis; [statistical method as in outcome 1, analysis 3]

13. Secondary Outcome: Self-perception of Body Attractiveness Assessed by Children and Youth Physical Self-perception Profile (CY-PSPP)
Description: The scale "Children and Youth Physical Self Perception Profile (CY-PSPP)" assessed the children's self-percetion about body attractiveness subscale in both groups at the beginning and at the end of protocol. The subscale was assessed by 6 questions with four ordinal levels (1-4) of response. Minimum and maximum total scores change between 6 to 24 for the subscale. Higher scores mean a better score.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
score on a scale
  At the beginning of games | 17.37 (2.78) | 16.11 (3.17)
  At the end of the games | 18.69 (3.57) | 17.11 (4.19)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable self-perception of body attractiveness; Test type: Superiority; p = 0.638505, ANCOVA — The outcome of self-perception for body attractiveness was tested for any difference between groups by covariate analysis; Adjusted for self-perception for body attractiveness at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.632, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; Adjusted for cluster effect in addition to baseline value and age
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.63280, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

14. Secondary Outcome: Self-perception of Global Physical Self-worth Assessed by Children and Youth Physical Self-perception Profile (CY-PSPP)
Description: The scale "Children and Youth Physical Self Perception Profile (CY-PSPP)" assessed the children's self-percetion about physical self-worth subscale in both groups at the beginning and at the end of protocol. The subscale was assessed by 6 questions with four ordinal levels (1-4) of response. Minimum and maximum total scores change between 6 to 24 for the subscale. Higher scores mean a better score.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
score on a scale
  At the beginning of games | 18.03 (2.50) | 17.37 (2.74)
  At the end of the games | 20.32 (2.48) | 18.15 (4.05)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable self-perception of global physical self-worth; Test type: Superiority; p = 0.007061, ANCOVA — The outcome of self-perception of global physical self-worth was tested for any difference between groups by covariate analysis; Adjusted for self-perception for global physical self-worth at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.005, Linear mixed effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.00603, Linear mixed-effects model — Linear mixed-effects model fit by maximum likelihood since restricted maximum likelihood assumes a strong normality; [statistical method as in outcome 1, analysis 3]

15. Secondary Outcome: Self-perception of Global Self-worth Assessed by Children and Youth Physical Self-perception Profile (CY-PSPP)
Description: The scale "Children and Youth Physical Self Perception Profile (CY-PSPP)" assessed the children's self-percetion about global self-worth subscale in both groups at the beginning and at the end of protocol. The subscale was assessed by 6 questions with four ordinal levels (1-4) of response. Minimum and maximum total scores change between 6 to 24 for the subscale. Higher scores mean a better score.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 53 | 53
score on a scale
  At the beginning of games | 18.03 (2.50) | 17.92 (2.65)
  At the end of the games | 20.69 (2.80) | 18.69 (4.25)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Null hypothesis was the absence of difference between the two groups for the dependent variable self-perception of global self-worth; Test type: Superiority; p = 0.002879, ANCOVA — The outcome of self-perception for global self-worth was tested for any difference between groups by covariate analysis; Adjusted for self-perception for global self-worth at baseline and confounding variable age
Statistical Analysis 2: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.002, Linear mixed effects model — [p-value comment as in outcome 10, analysis 3]; [statistical method as in outcome 1, analysis 3]
Statistical Analysis 3: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.00238, Linear mixed-effects model — [p-value comment as in outcome 10, analysis 3]; [statistical method as in outcome 1, analysis 3]

16. Secondary Outcome: Enjoyment Levels of Genders From Sports Category in the Game Group by Physical Activity Enjoyment Scale (PACES-SF)
Description: For Sports category, there were 5 games of boxing, tennis, golf, baseball, and bowling. Thus, each child was evaluated after every single game by five bipolar scale questions. Questions 1 and 4 were starting from positive to negative answers (left to right) and scored as 7-1. Scale scores were determined by calculating the mean. All scale scores were summed to calculate the Category score. The higher the score, the better the enjoyment in this category.
  Min-Max Sports Category scores were 11-25 for females and 17.8-26.2 for males.
Time Frame: After every game during 12 weeks
Population: Enjoyment levels only in the intervention group were assessed since control group did not play the games of interest.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Female: Females' enjoyment levels in AVG group playing Nintendo Wii® active video game categories of sports (boxing, tennis, golf, baseball, and bowling), balance (ski slalom, heading ball, balance bubble, ski jumping and penguin playing), aerobics (rhythm boxing,hula-hoop, cycling, step, and run), resort (jet-skiing, water skiing, table tennis, basketball, swordplay, archery, canoeing and frisbee) and training (rhythm kung fu, snowball, turning ball, Segway circuit, perfect 10, skateboard, major, obstacle course and bicycle).
- Males: Males' enjoyment levels in AVG group playing Nintendo Wii® active video game categories of sports (boxing, tennis, golf, baseball, and bowling), balance (ski slalom, heading ball, balance bubble, ski jumping and penguin playing), aerobics (rhythm boxing,hula-hoop, cycling, step, and run), resort (jet-skiing, water skiing, table tennis, basketball, swordplay, archery, canoeing and frisbee) and training (rhythm kung fu, snowball, turning ball, Segway circuit, perfect 10, skateboard, major, obstacle course and bicycle).
Arm/Group | Female | Males
Number analyzed (Participants) | 29 | 24
score on a scale | 21.34 (2.59) | 20.46 (4.08)
Statistical Analysis 1: Comparison: Female vs Males; Enjoyment scale of physical activity "sports" in intervention group between male and female genders; Test type: Superiority; p = 0.194, Wilcoxon (Mann-Whitney) — Tested the significance of gender between genders

17. Secondary Outcome: Enjoyment Levels of Genders From Resort Category in the Game Group by Physical Activity
Description: For Resort category, there were 8 games of jet-skiing, water skiing, table tennis, basketball, swordplay, archery, canoeing and frisbee. Thus, each child was evaluated after every single game by five bipolar scale questions. Questions 1 and 4 were starting from positive to negative answers (left to right) and therefore scored as 7-1. Scale scores were determined by calculating the mean. All scale scores were summed to calculate the Category score. The higher the score, the better the enjoyment in this category.
  Min-Max Resort Category scores were 23.2-37 for females and 25.8-37.8 for males.
Time Frame: After every game during 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Female: Females' enjoyment levels in AVG group playing Nintendo Wii® active video game categories of resort (jet-skiing, water skiing, table tennis, basketball, swordplay, archery, canoeing and frisbee).
- Males: Males' enjoyment levels in AVG group playing Nintendo Wii® active video game categories of resort (jet-skiing, water skiing, table tennis, basketball, swordplay, archery, canoeing and frisbee).
Arm/Group | Female | Males
Number analyzed (Participants) | 29 | 24
score on a scale | 33.04 (3.36) | 33.27 (3.30)
Statistical Analysis 1: Comparison: Female vs Males; Null hypothesis was the absence of difference between the two genders in the Active video game group for the variable of enjoyment from sports category; Test type: Superiority; p = 0.809, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Enjoyment Levels by Physical Activity of Genders From Balance Category in the Game Group
Description: For Balance category, there were 5 games of ski slalom, heading ball, balance bubble, ski jumping and penguin playing. Thus, each child was evaluated after every single game by five bipolar scale questions. Questions 1 and 4 were starting from positive to negative answers (left to right) and therefore scored as 7-1. Scale scores were determined by calculating the mean. All scale scores were summed to calculate the Category score. The higher the score, the better the enjoyment in this category.
  Min-Max Balance Category scores were 14.4-23.2 for females and 15-26.6 for males.
Time Frame: After every game during 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Female: Females' enjoyment levels in AVG group playing Nintendo Wii® active video game categories of balance (ski slalom, heading ball, balance bubble, ski jumping and penguin playing).
- Males: Males' enjoyment levels in AVG group playing Nintendo Wii® active video game categories of balance (ski slalom, heading ball, balance bubble, ski jumping and penguin playing).
Arm/Group | Female | Males
Number analyzed (Participants) | 29 | 24
score on a scale | 21.24 (2.32) | 21.41 (2.49)
Statistical Analysis 1: Comparison: Female vs Males; Null hypothesis was the absence of difference between the two genders in the active video game group for the variable of enjoyment from balance category; Test type: Superiority; p = 0.843, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Enjoyment Levels by Physical Activity of Genders From Aerobic Category in the Game Group
Description: For Aerobics category, there were 5 games of rhytmic boxing, hula-hoop, cycling, step, and run. Thus, each child was evaluated after every single game by five bipolar scale questions. Questions 1 and 4 were starting from positive to negative answers (left to right) and therefore scored as 7-1. Scale scores were determined by calculating the mean. All scale scores were summed to calculate the Category score. The higher the score, the better the enjoyment in this category.
  Min-Max Aerobics Category scores were 17.8-24 for females and 14.4-26.4 for males.
Time Frame: After every game during 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Female: Females' enjoyment levels in AVG group playing Nintendo Wii® active video game category of aerobics (rhythm boxing,hula-hoop, cycling, step, and run).
- Males: Males' enjoyment levels in AVG group playing Nintendo Wii® active video game category of aerobics (rhythm boxing,hula-hoop, cycling, step, and run).
Arm/Group | Female | Males
Number analyzed (Participants) | 29 | 24
score on a scale | 22.17 (1.41) | 21.54 (2.39)
Statistical Analysis 1: Comparison: Female vs Males; Null hypothesis was the absence of difference between the two genders in the active video game group for the variable of enjoyment from aerobic category; Test type: Superiority; p = 0.247, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Enjoyment Levels by Physical Activity of Genders From Training Category in the Game Group
Description: For Training category, there were 9 games of rhythm kung fu, snowball, turning ball, Segway circuit, perfect 10, skateboard, major, obstacle course and bicycle. Thus, each child was evaluated after every single game by five bipolar scale questions. Questions 1 and 4 were starting from positive to negative answers (left to right) and therefore scored as 7-1. Scale scores were determined by calculating the mean. All scale scores were summed to calculate the Category score. The higher the score, the better the enjoyment in this category.
  Min-Max Training Category scores were 31.6-41.8 for females and 29.2-45.2 for males.
Time Frame: After every game during 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Female: Females' enjoyment levels in AVG group playing Nintendo Wii® active video game categories of training (rhythm kung fu, snowball, turning ball, Segway circuit, perfect 10, skateboard, major, obstacle course and bicycle).
- Males: Males' enjoyment levels in AVG group playing Nintendo Wii® active video game categories of training (rhythm kung fu, snowball, turning ball, Segway circuit, perfect 10, skateboard, major, obstacle course and bicycle).
Arm/Group | Female | Males
Number analyzed (Participants) | 29 | 24
score on a scale | 38.50 (2.70) | 37.95 (3.61)
Statistical Analysis 1: Comparison: Female vs Males; Null hypothesis was the absence of difference between the two genders in the active video game group for the variable of enjoyment from training category; Test type: Superiority; p = 0.543, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53

LIMITATIONS AND CAVEATS:
Conforming strictly to the rules of CONSORT extension for such "well controlled" studies when clustering with huge numbers of clusters without the risk of contamination might be impossible and unnecessary in small research areas like the city, Bolu.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes